CLINICAL TRIAL: NCT00463684
Title: Assessment of the Immunogenicity and Safety of Japanese Encephalitis Live Attenuated SA 14-14-2 Vaccine in Children in Sri Lanka
Brief Title: Live Attenuated Japanese Encephalitis (JE) Vaccine Coadministered With Measles Vaccine in Infants 9 Months of Age
Acronym: JEV03
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Ministry of Health of Sri Lanka (Unknown); Mahidol University (Other); Quintiles Singapore (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JEV03
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): Healthy infants 9 months of age (plus or minus 2 weeks) that met the eligibility criteria. Subjects received one dose of Live, Attenuated Japanese Encephalitis SA 14-14-2 Vaccine (LJEV) and one dose of live, attenuated measles vaccine.
  Interventions: Biological: Live, Attenuated Japanese Encephalitis SA 14-14-2 Vaccine; Biological: Live, attenuated measles vaccine

INTERVENTIONS:
Biological: Live, Attenuated Japanese Encephalitis SA 14-14-2 Vaccine — Manufactured by Chengdu Institute of Biological Products (CDIBP), Chengdu, China; batch 200611A078-1. Administered subcutaneously in the right brachium.
Biological: Live, attenuated measles vaccine — Manufactured by Serum Institute of India, Ltd, Pune, India; batch EU3244. Administered subcutaneously in the left brachium.

SUMMARY:
To facilitate introduction of live attenuated SA 14-14-2 Japanese encephalitis vaccine (LJEV) into the National Immunization Programme of Sri Lanka, we evaluated the safety and immunogenicity of co-administration of LJEV and measles vaccine at 9 months of age. The primary hypothesis was that the seropositivity rate at 28 days post vaccination in Japanese Encephalitis (JE) and measles concomitantly vaccinated subjects 9 months of age is greater than 80% for JE and greater than 90% for measles.

DETAILED DESCRIPTION:
JE virus is an arbovirus that causes a devastating neurological disease resulting in high rates of mortality orneurologic sequelae. The severity of sequelae, together with the volume of cases, makes JE an important cause of encephalitis. The disease is endemic across temperate and tropical zones of Asia,and because of its zoonotic cycle, eradicating JE from the environment is unrealistic. Universal childhood vaccination is essential for disease control. In Sri Lanka, immunization against JE began in 1988. By 2006, two types of JE vaccines were available for use in Sri Lanka-inactivated mouse brain-derived vaccine and live attenuated SA-14-14-2 JE vaccine (LJEV). Only the inactivated vaccine was being used in the country's public-sector immunization program. Concern in Japan over a rare but potentially dangerous adverse event associated with a mouse brain-derived vaccine led the manufacturer in Japan to discontinue production in 2005, thus limiting global supply of inactivated JE vaccines and raising costs for remaining inactivated vaccines. In August of 2006, the World Health Organization stated in its position paper on Japanese encephalitis vaccines that the mouse brain-derived vaccine should be replaced by a new generation of JE vaccines. For Sri Lanka, switching to the less expensive LJEV was estimated in 2006 to save the National Immunization Programme (NIP) between US$8.6 and $8.9 million annually in direct vaccine costs alone. To generate local immunogenicity and safety data to guide policy for potential use of LJEV in Sri Lanka's NIP, the Ministry of Healthcare and Nutrition, in cooperation with PATH, initiated the study. The study was conducted in three peri-urban health divisions of low JE endemicity in the District of Colombo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy child 9 months (±2 weeks) of age at the enrollment visit.
* Subject was a full-term infant.
* Subject's parent or legal guardian is literate and willing to provide written informed consent.
* Subject is up-to-date for all vaccinations recommended in the Sri Lankan childhood immunization schedule.

Exclusion Criteria:

* Enrolled in another clinical trial involving any therapy.
* Subject and/or parent(s) or guardian(s) are unable to attend the scheduled visits or comply with the study procedures.
* Received any non-study vaccine within 2 weeks prior to enrolment or refusal to postpone receipt of such vaccines until 28 days after study entry.
* Prior or anticipated receipt of immune globulin or other blood products, or injected or oral corticosteroids or other immune modulator therapy except routine vaccines within 6 weeks of administration of study vaccine. Individuals on a tapering dose schedule of oral steroids lasting <7 days may be included in the trial as long as they have not received more than one course within the last 2 weeks prior to enrolment.
* History of documented or suspected encephalitis, encephalopathy, or meningitis.
* History of measles.
* History of Japanese encephalitis.
* Serious adverse event related (i.e., possible, probably, definite) to previous receipt of any JE vaccine, if applicable.
* Persistent inconsolable crying (>3 hours) observed after previous receipt of any JE vaccine, if applicable.
* Hypotonic - hyporesponsiveness after past receipt of any JE vaccine, if applicable.
* Suspected or known hypersensitivity to any of the investigational or marketed vaccine components.
* History of serious chronic disease (cardiac, renal, neurologic, metabolic, or rheumatologic).
* Underlying medical condition such as inborn errors of metabolism, failure to thrive, bronchopulmonary dysplasia, or any major congenital abnormalities requiring surgery or chronic treatment.
* History of thrombocytopenic purpura.
* History of seizures, including history of febrile seizures, or any other neurologic disorder.
* Known or suspected immunologic function impairment of any kind and/or known HIV infection.
* Parent with known or suspected immunologic function impairment of any kind and/or known HIV infection.
* Any condition that, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the study objectives.

Ages: 9 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2007-07-07; Primary Completion 2007-11-07 (Actual); Study Completion 2008-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Abeysinghe, MD, MSc, Principal Investigator — Epidemiological Unit, Sri Lanka Ministry of Healthcare and Nutrition
Locations (3):
- Sri Lanka (3):
  - Homagama MOH Division Medical Office, Homagama, District of Colombo
  - Kolonnawa MOH Division Medical Office, Kolonnawa, District of Colombo
  - Moratuwa MOH Division Medical Office, Moratuwa, District of Colombo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subject children were identified through Ministry of Health (MOH) birth and immunization registries of selected vaccination clinics.
Period: Overall Study
Arm/Group | All Subjects
Started | 278
Completed | 274
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 278
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.2 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 130
Region of Enrollment [Number; unit: participants]
  Sri Lanka | 278

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With Demonstrated Seropositivity for Japanese Encephalitis (JE) Neutralizing Antibodies
Description: Blood serum was collected immediately before administration (Day 0), Day 28, six months post-administration, and 1 year later. Serum neutralizing antibodies to the Beijing-1 JE strain were measured by plaque reduction neutralization test (PRNT) where the neutralizing titer was measured as the inverse dilution at which plaque counts were reduced by 50%. Seropositivity was defined as a titer of ≥1:10.
Time Frame: 1 year
Population: Of the 278 enrolled, 257 participants were determined to meet criteria at 28 days weeks post-co-administration with study vaccines (13 were found to have been out of range for age at inclusion, 4 did not have the Day 28 blood specimen collected within range, and 4 were not able to provide sera at Day 28).
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 257
Participants
  Day 0: Yes | 14
  Day 0: No | 243
  Day 28: Yes | 233
  Day 28: No | 24
  6 months: number analyzed (Participants) | 243
  6 months: Yes | 202
  6 months: No | 41
  1 year: number analyzed (Participants) | 253
  1 year: Yes | 221
  1 year: No | 32

2. Primary Outcome: Number and Percentage of Subjects With Demonstrated Seropositivity for Anti-measles Immunoglobulin G (IgG): Manufacturer Definition
Description: Blood serum was collected immediately before administration (Day 0), Day 28, six months post-administration, and 1 year later. Serum anti-measles immunoglobulin class G (IgG) antibodies were measured by enzyme-linked immunosorbent assay (ELISA) (Serion ELISA classic Measles Virus IgG, Serion GmbH, Würzburg,Germany). For anti-measles IgG, two definitions of seropositivity were used: per manufacturer's instruction (concentration of>200 mIU/mL, this table) and when including those with "borderline" results (≥150 mIU/mL).
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 257
Participants
  Day 0: Yes | 0
  Day 0: No | 257
  Day 28: Yes | 218
  Day 28: No | 39
  6 months: number analyzed (Participants) | 243
  6 months: Yes | 229
  6 months: No | 14
  1 year: number analyzed (Participants) | 253
  1 year: Yes | 246
  1 year: No | 7

3. Primary Outcome: Number and Percentage of Subjects With Demonstrated Seropositivity for Anti-measles Immunoglobulin G (IgG): Including Borderline Subjects
Description: Blood serum was collected immediately before administration (Day 0), Day 28, six months post-administration, and 1 year later. Serum anti-measles immunoglobulin class G (IgG) antibodies were measured by enzyme-linked immunosorbent assay (ELISA) (Serion ELISA classic Measles Virus IgG, Serion GmbH, Würzburg,Germany). For anti-measles IgG, two definitions of seropositivity were used: per manufacturer's instruction (concentration of>200 mIU/mL) and when including those with "borderline" results (≥150 mIU/mL, this table).
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 257
Participants
  Day 0: Yes | 0
  Day 0: No | 257
  Day 28: Yes | 244
  Day 28: No | 13
  6 months: number analyzed (Participants) | 243
  6 months: Yes | 229
  6 months: No | 14
  1 year: number analyzed (Participants) | 253
  1 year: Yes | 246
  1 year: No | 7

4. Secondary Outcome: Geometric Mean Titer (GMT) of Japanese Encephalitis (JE) Neutralizing Antibodies
Description: Blood serum was collected immediately before administration (Day 0), Day 28, six months post-administration, and 1 year later. Serum neutralizing antibodies to the Beijing-1 JE strain were measured by plaque reduction neutralization test (PRNT) where the neutralizing titer was measured as the inverse dilution at which plaque counts were reduced by 50%.
Time Frame: 1 year
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | All Subjects
Number analyzed (Participants) | 257
titer
  Day 0 | 5.5 [5.2 to 5.8]
  Day 28 | 110.6 [90.3 to 135.4]
  6 months: number analyzed (Participants) | 243
  6 months | 68.3 [55.3 to 83.4]
  1 year: number analyzed (Participants) | 253
  1 year | 75.5 [62.2 to 91.6]

5. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-measles Immunoglobulin G (IgG)
Description: as for outcome 2
Time Frame: 1 year
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | All Subjects
Number analyzed (Participants) | 257
titer
  Day 0 | 20.5 [18.4 to 22.8]
  Day 28 | 374.9 [351.0 to 400.4]
  6 months | 697.8 [634.0 to 768.0]
  1 year | 1201.7 [1076.7 to 1341.3]

6. Secondary Outcome: Number and Percentage of Subjects With Immediate Reactions, Local and Systemic Reactions, and Unsolicited Adverse Events (AE)
Description: Subjects were monitored for immediate AEs and local reactions for 30 minutes after each injection by a study physician. Thereafter, parents recorded axillary temperature, local reactions (redness, swelling, pain, and other local reactions), and systemic symptoms (high-grade fever, anorexia, crying, diarrhea, drowsiness, insomnia, irritability, vomiting, and other systemic symptoms) in a study diary for 7 days afterwards. Study staff called the subjects' parents 2 days after vaccination and monthly through 1 year to inquire about the child's well being and review the diary card. The subject was visited at home on Day 7 to review and collect the reactogenicity diary card. The subject returned to the vaccination clinic on Day 28, 6 months, and 1 year to be examined, have a blood draw, and review any AEs or serious adverse events (SAE) with parents.
Time Frame: 1 year
Population: Not all subjects were followed for a full 30 minutes after injection.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 278
Participants
  Immediate reaction: number analyzed (Participants) | 254
  Immediate reaction: Yes | 0
  Immediate reaction: No | 254
  Solicited local reaction: LJEV, Days 0-3: Yes | 34
  Solicited local reaction: LJEV, Days 0-3: No | 244
  Solicited local reaction: measles, Days 0-3: Yes | 27
  Solicited local reaction: measles, Days 0-3: No | 251
  Solicited local reactions, LJEV: Days 4-7: Yes | 2
  Solicited local reactions, LJEV: Days 4-7: No | 276
  Solicited local reactions, measles: Days 4-7: Yes | 1
  Solicited local reactions, measles: Days 4-7: No | 277
  Solicited systemic reaction, days 0-7: Yes | 112
  Solicited systemic reaction, days 0-7: No | 166
  Solicited systemic reaction, >7 days: Yes | 18
  Solicited systemic reaction, >7 days: No | 260
  Unsolicited systemic reactions, Days 0-7: Yes | 30
  Unsolicited systemic reactions, Days 0-7: No | 248
  Unsolicited systemic reactions, >7 days: Yes | 14
  Unsolicited systemic reactions, >7 days: No | 264
  Any non-serious adverse event: Yes | 122
  Any non-serious adverse event: No | 156
  Related adverse events: Yes | 0
  Related adverse events: No | 278
  Serious adverse events, Days 8-365: Yes | 45
  Serious adverse events, Days 8-365: No | 233

7. Secondary Outcome: Number of Solicited Local Reactions to LJEV: Days 0-3
Description: Parents recorded axillary temperature, local reactions (redness, swelling, pain, and other local reactions), and systemic symptoms (high-grade fever, anorexia, crying, diarrhea, drowsiness, insomnia, irritability, vomiting, and other systemic symptoms) in a study diary for 7 days after vaccination. The subject was visited at home on Day 7 to review and collect the reactogenicity diary card.
Time Frame: 3 days
Measure: Number; unit: reactions
Arm/Group | All Subjects
Number analyzed (Participants) | 278
reactions
  Any solicited local reaction: Any severity | 34
  Any solicited local reaction: Grade 3 | 0
  Erythema: Any severity | 11
  Erythema: Grade 3 | 0
  Induration: Any severity | 7
  Induration: Grade 3 | 0
  Pain: Any severity | 25
  Pain: Grade 3 | 0

8. Secondary Outcome: Number of Solicited Local Reactions to LJEV: Days 4-7
Description: as for outcome 7
Time Frame: 4 days
Measure: Number; unit: reactions
Arm/Group | All Subjects
Number analyzed (Participants) | 278
reactions
  Any solicited local reaction: Any severity | 2
  Any solicited local reaction: Grade 3 | 0
  Erythema: Any severity | 1
  Erythema: Grade 3 | 0
  Induration: Any severity | 0
  Induration: Grade 3 | 0
  Pain: Any severity | 1
  Pain: Grade 3 | 0

9. Secondary Outcome: Number of Solicited Local Reactions to Measles Vaccine: Days 0-3
Description: as for outcome 7
Time Frame: 3 days
Measure: Number; unit: reactions
Arm/Group | All Subjects
Number analyzed (Participants) | 278
reactions
  Any solicited local reaction: Any severity | 27
  Any solicited local reaction: Grade 3 | 0
  Erythema: Any severity | 11
  Erythema: Grade 3 | 0
  Induration: Any severity | 6
  Induration: Grade 3 | 0
  Pain: Any severity | 21
  Pain: Grade 3 | 0

10. Secondary Outcome: Number of Solicited Local Reactions to Measles Vaccine: Days 4-7
Description: as for outcome 7
Time Frame: 4 days
Measure: Number; unit: reactions
Arm/Group | All Subjects
Number analyzed (Participants) | 278
reactions
  Any solicited local reaction: Any severity | 1
  Any solicited local reaction: Grade 3 | 0
  Erythema: Any severity | 1
  Erythema: Grade 3 | 0
  Induration: Any severity | 0
  Induration: Grade 3 | 0
  Pain: Any severity | 0
  Pain: Grade 3 | 0

11. Secondary Outcome: Number of Solicited Systemic Reactions: Days 0-3
Description: as for outcome 7
Time Frame: 3 days
Measure: Number; unit: reactions
Arm/Group | All Subjects
Number analyzed (Participants) | 278
reactions
  Any solicited systemic reaction: Any severity | 105
  Any solicited systemic reaction: Grade 3 | 4
  Fever: Any severity | 21
  Fever: Grade 3 | 0
  Anorexia: Any severity | 52
  Anorexia: Grade 3 | 0
  Crying: Any severity | 56
  Crying: Grade 3 | 0
  Diarrhea: any severity | 27
  Diarrhea: Grade 3 | 2
  Tiredness: Any severity | 32
  Tiredness: Grade 3 | 0
  Insomnia: Any severity | 33
  Insomnia: Grade 3 | 1
  Irritability: Any severity | 17
  Irritability: Grade 3 | 0
  Vomiting: Any severity | 17
  Vomiting: Grade 3 | 1

12. Secondary Outcome: Number of Solicited Systemic Reactions: Days 4-7
Description: as for outcome 7
Time Frame: 4 days
Measure: Number; unit: reactions
Arm/Group | All Subjects
Number analyzed (Participants) | 278
reactions
  Any solicited systemic reaction: Any severity | 55
  Any solicited systemic reaction: Grade 3 | 2
  Fever: Any severity | 14
  Fever: Grade 3 | 0
  Anorexia: Any severity | 32
  Anorexia: Grade 3 | 0
  Crying: Any severity | 18
  Crying: Grade 3 | 0
  Diarrhea: any severity | 19
  Diarrhea: Grade 3 | 2
  Tiredness: Any severity | 11
  Tiredness: Grade 3 | 0
  Insomnia: Any severity | 15
  Insomnia: Grade 3 | 0
  Irritability: Any severity | 10
  Irritability: Grade 3 | 0
  Vomiting: Any severity | 6
  Vomiting: Grade 3 | 0

ADVERSE EVENTS:
Time Frame: 1 year for serious adverse events, 28 days for non-serious adverse events.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/278
Serious Adverse Events (participants affected / at risk) | 45/278
Other Adverse Events (participants affected / at risk) | 122/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=278)
Conjunctivitis (Eye disorders) | 1 (1)
Anal skin tags (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Dysentery (Infections and infestations) | 1 (1)
Eczema infected (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 11 (13)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 7 (7)
Otitis media acute (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 8 (9)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Febrile convulsion (Nervous system disorders) | 3 (4)
Genital labial adhesions (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=278)
Conjunctivitis (Eye disorders) | 1 (1)
Anal skin tags (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (13)
Vomiting (Gastrointestinal disorders) | 8 (9)
Gait disturbance (Gastrointestinal disorders) | 1 (1)
Pyrexia (Gastrointestinal disorders) | 38 (39)
Food allergy (Immune system disorders) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Dysentery (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1 (1)
Eczema infected (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 11 (12)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 10 (10)
Nasopharyngitis (Infections and infestations) | 34 (35)
Otitis media acute (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 8 (9)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Febrile convulsion (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 1 (1)
Crying (Psychiatric disorders) | 1 (1)
Genital labial adhesions (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (46)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No